CLINICAL TRIAL: NCT05884710
Title: Effectıveness of Foot Core Exercises on paın and functıonal Performance ın patıents wıth Patellofemoral paın Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 777
Record Dates: First submitted 2023-05-09; First posted 2023-06-01 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Intervention Model Description: Participants with Patellofemoral Pain Syndrome (PFPS) will be randomly divided into 2 groups.
Who Masked: Participant
Masking Description: 30 participants with patellofemoral pain syndrome
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): Foot core exercises consist of 4 movements; short foot exercise, towel curls, toe spread and squeeze, balance board training
  Interventions: Other: Foot core exercises; Other: Conventional Physiotherapy
- Control Group (Active Comparator): Conventional Physiotherapy Program
  Interventions: Other: Conventional Physiotherapy

INTERVENTIONS:
Other: Foot core exercises — 2 groups; First group is an intervention group who has contain foot core exercises and the other group is a control group.
  Arms: Exercise Group
Other: Conventional Physiotherapy — Electrotherapeutic modalities and range of motion exercises

SUMMARY:
30 participants wit Patellofemoral Pain Syndrome will be included in this study.Participants will be randomly divided and divided into 2 groups: The first group contains; quadrıceps ısometrıc exercıses ın supıne posıtıon, NMES electrıcal current, soft tıssue therapy-patellar mobılısatıon and the second group contains:quadrıceps ısometrıc exercıses ın supıne posıtıon, NMES electrıcal current, soft tıssue therapy-patellar mobılısatıon and foot core exercıses (short foot exercise, towel curls, toe spread and squeeze, balance board training).

DETAILED DESCRIPTION:
This study will be carried out in Mersin Medikalpark Hospital and this research planned as a prospective, randomized controlled trial.30 participants with Patellofemoral Pain Syndrome (PFPS) will be included in this study.Some inclusion and exclusion criterias were determined for our study.İnclusion criterias are volunteering to participate in research,participants between 20-59 years old with PFPS will be included if they had anterior knee pain during at least 2 funtional activities including step-up and step-down, squatting,kneeling,jumping or running of at least 1 months' duration,individuals who are active for 30 minutes almost every day of the week,individuals who has with chondromalacia patella grade 1-2-3 and lateral patellar compression syndrome.Exclusion criterias are acute musculoskeletal injury affecting the lower extremity in the last 4 months, having a balance or vestibular disorder,low quality of life,limited lower extremity movements.Participants will be randomly divided and divided into 2 groups: The first group contains; quadrıceps ısometrıc exercıses ın supıne posıtıon, NMES electrıcal current, soft tıssue therapy-patellar mobılısatıon and the second group contains:quadrıceps ısometrıc exercıses ın supıne posıtıon, NMES electrıcal current, soft tıssue therapy-patellar mobılısatıon and foot core exercıses (short foot exercise, towel curls, toe spread and squeeze, balance board training).Some measurement parameters will be used in this study. VAS scale will be used to assess pain.10 meter walk test,timed up and go test, stair climb test and Internatıonal Physical Actıvıty Questionnaire(IPAQ) will be used to assess functional performance.Knee and ankle muscle test and range of motions will assessed and quality of life will evaluated with SF-36 short form scale.All measurements will be made again after 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* İnclusion criterias are volunteering to participate in research,participants between 20-59 years old with PFPS will be included if they had anterior knee pain during at least 2 funtional activities including step-up and step-down, squatting,kneeling,jumping or running of at least 1 months' duration,individuals who are active for 30 minutes almost every day of the week,individuals who has with chondromalacia patella grade 1-2-3 and lateral patellar compression syndrome

Exclusion Criteria:

* Exclusion criterias are acute musculoskeletal injury affecting the lower extremity in the last 4 months,having a balance or vestibular disorder,low quality of life,limited lower extremity movements.

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | 6 weeks
  The scale called VAS will be used for pain assessment. Patirnt will select the number between 0 and 10. While 0 means no pain, 10 means worst pain.
10 meter walk test | 6 weeks
  Walking test for assess functional performance
Timed up and go test | 6 weeks
  Walking test for assess functional performance
Stair climb test | 6 weeks
  Step in and out for assess functional performance
International Physical Activity Questionnaire | 6 weeks
  This is a scale for functional performance

SECONDARY OUTCOMES:
SF-36 short form | 6 weeks
  Quality of life
Knee and ankle ROM | 6 weeks
  Knee and ankle range of motion values

CONTACTS AND LOCATIONS:
Locations (1):
- Yeditepe University, Istanbul, İnönü Mah. Kayışdağı Cad. 326a. 26 Ağustos Yerleşimi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No